CLINICAL TRIAL: NCT02595554
Title: Neoadjuvant Chemotherapy and Radical Surgery Versus Concurrent Chemoirradiation in FIGO Stage IIB Cervical Cancer
Brief Title: Neoadjuvant Chemotherapy and Radical Surgery in Stage IIB Cervical Cancer
Acronym: SYSGO002
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSEM007
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Cervical Carcinoma Stage IIB
Keywords: Cervical cancer, Stage IIB, Neoadjuvant chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Surgical Procedures, Operative; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoirradiation (CCRT) (Active Comparator): Concurrent chemoirradiation
  Interventions: Radiation: Concurrent chemoirradiation
- NACT+Surgery (Experimental): Neoadjuvant chemotherapy with Paclitaxel and Cisplatin (3 cycles), followed by radical surgery
  Interventions: Drug: Paclitaxel; Procedure: Radical Surgery; Drug: Cisplatin

INTERVENTIONS:
Radiation: Concurrent chemoirradiation — External beam radiation therapy (EBRT) with concurrent weekly platinum chemotherapy followed by brachytherapy
  Arms: Concurrent chemoirradiation (CCRT)
Drug: Paclitaxel — New adjuvant chemotherapy 3 cycles with Paclitaxel 150mg/m2 over 3 hours and Cisplatin
  Other Names: NACT
  Arms: NACT+Surgery
Procedure: Radical Surgery — Radical hysterectomy (Type III or Type IV hysterectomy) plus bilateral pelvic lymph node dissection and para-aortic lymph node dissection or sampling
  Other Names: NACT and surgery
  Arms: NACT+Surgery
Drug: Cisplatin — New adjuvant chemotherapy 3 cycles with Paclitaxel and Cisplatin 70mg/m2
  Other Names: NACT
  Arms: NACT+Surgery

SUMMARY:
Neoadjuvant chemotherapy (NACT) and radical surgery (RS) may have a possible better outcome to concurrent chemoirradiation (CCRT) in stage IIB cervical cancer. We try to verify such a hypothesis in terms of survival and treatment related morbidity.

DETAILED DESCRIPTION:
Patients with International Federation of Gynecology and Obstetrics (FIGO) stage IIB cervical cancer are eligible for our study. They will receive cisplatin based neoadjuvant chemotherapy (NACT) 3 cycles followed by radical surgery (RS) (type III to V radical hysterectomy plus systematic pelvic lymphadenectomy) (arm A) or external beam radiation (EBRT) with concurrent weekly platinum 40mg/m2 followed by brachyradiotherapy (arm B).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed cervical carcinoma
* Original clinical stage must be IIB （FIGO 2009）
* Histopathology squamous carcinoma, adenocarcinoma or adeno-squamous carcinoma
* Age between 18-65
* Patients must give signed informed consent

Exclusion Criteria:

* The presence of uncontrolled life-threatening illness
* Receiving other ways of anti-cancer therapy
* Investigator consider the patients can't finish the whole study
* With normal liver function test (ALT、AST>2.5×ULN)
* With normal renal function test (Creatinine>1.5×ULN)
* WBC<4,000/mm3 or PLT<100,000/mm3

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph. D, Study Director — Sun Yat-sen University
Locations (1):
- Department of Gynecologic Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tu H, Huang H, Ouyang Y, Liu Q, Xian B, Song K, Chen G, Shen Y, Liu J. Neoadjuvant chemotherapy followed by radical surgery versus concurrent chemoradiotherapy in patients with FIGO stage IIB cervical cancer: the CSEM 006 study. Int J Gynecol Cancer. 2021 Jan;31(1):129-133. doi: 10.1136/ijgc-2020-001357. Epub 2020 Jun 9. PMID 32522771